CLINICAL TRIAL: NCT00924105
Title: A Two-Stage Randomized Placebo-controlled Ascending Dose Phase I/ IIa Study to Evaluate Safety, Tolerability, Pharmacodynamic Effects and Preliminary Efficacy of an Anti-Interleukin 1 Beta Vaccine (CYT013-IL1bQb) in Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability and Pharmacodynamics of CYT013-IL1bQb in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYT013-IL1bQb 01
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CYT013-IL1bQb
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CYT013-IL1bQb — s.c. injection
  Arms: 1
Drug: Placebo — s.c. injection
  Arms: 2

SUMMARY:
The purpose of this clinical trial is to test safety and tolerability of a vaccine targeting Interleukin-1 beta in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus, according to the American Diabetes Association diagnostic criteria, ≥ 3 months at time of randomization
* HbA1c in the range of 6.5 - 9.5% (inclusive) at screening
* Treatment with diet and exercise alone or a stable dose of metformin, or sulfonylurea, or metformin plus a sulfonylurea for at least 4 weeks prior to randomization
* Further criteria as defined in the clinical trial protocol

Exclusion Criteria:

* Symptoms of hyperglycemia (i.e. polyuria and polydypsia)
* History of significant weight gain or loss (+/-5%) during the 4 weeks before randomization
* Fasting C-peptide level < 400 pmol/L at screening
* Change in the medicamentous treatment of elevated blood pressure, diabetes mellitus or dyslipidemia within 4 weeks prior to the randomization
* Use of any weight loss medication (over the counter prescription) or initiation of a prescribed weight management or exercise program within 4 weeks before randomization
* Current systemic anti-inflammatory therapy other than aspirin ≤ 100 mg/day or immunosuppressive treatment, in particular oral corticosteroids

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | continously

SECONDARY OUTCOMES:
Biological measures of glycemia and inflammation | continously

CONTACTS AND LOCATIONS:
Locations (3):
- Cytos Investigator sites, Hamburg, Germany
- Switzerland (2):
  - Cytos Investigator sites, Basel
  - Cytos Investigator sites, Zurich

REFERENCES:
- [Derived] Cavelti-Weder C, Timper K, Seelig E, Keller C, Osranek M, Lassing U, Spohn G, Maurer P, Muller P, Jennings GT, Willers J, Saudan P, Donath MY, Bachmann MF. Development of an Interleukin-1beta Vaccine in Patients with Type 2 Diabetes. Mol Ther. 2016 May;24(5):1003-12. doi: 10.1038/mt.2015.227. Epub 2015 Dec 21. PMID 26686385